CLINICAL TRIAL: NCT06404528
Title: A Clinical Study on the Efficacy and Mechanism of Low-dose Chemotherapy Under Hypoglycaemia for the Treatment of Relapsed Refractory Advanced Solid Tumours
Brief Title: Low-dose Chemotherapy Under Hypoglycaemia for the Treatment of Relapsed Refractory Advanced Solid Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY23149
Record Dates: First submitted 2023-10-23; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumors, Adult
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood glucose stress combined with low-dose chemotherapy (Experimental): By controlling the patient's blood sugar, low-dose chemotherapy is used in a hypoglycemic state. Some necrotic tumor cells produced by chemotherapy can maintain their immunogenicity, further activate innate immunity, produce very strong anticancer effects, and have no cytotoxic reactions to chemotherapy.
  Interventions: Other: Blood glucose stress combined with low-dose chemotherapy

INTERVENTIONS:
Other: Blood glucose stress combined with low-dose chemotherapy — By controlling the patient's blood sugar, low-dose chemotherapy is used in a hypoglycemic state. Some necrotic tumor cells produced by chemotherapy can maintain their immunogenicity, further activate innate immunity, produce very strong anticancer effects, and have no cytotoxic reactions to chemotherapy.

SUMMARY:
By controlling the patient's blood sugar, small doses of chemotherapy are used in a hypoglycemic state. Some necrotic tumor cells produced by chemotherapy can maintain their immunogenicity, further activate innate immunity, and produce very strong anticancer effects without the cytotoxic effects of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years;
2. ASubjects must have histologically- or cytologically-confirmed diagnosis of advanced solid tumor(s) and have progressed on or is not eligible for available standard therapy;
3. Subjects have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
4. ECOG score of 0-2, lifespan > 12 weeks;
5. Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
6. Voluntarily participated in this study, signed the informed consent form, had good compliance, and cooperated with the follow-up

Exclusion Criteria:

1. The patient is diagnosed with central nervous system leukemia(symptoms, signs, imaging, cerebrospinal fluid);
2. White blood cell count ≥ 50×10^9/ L or patients with rapid disease progression can't be guaranteed to complete a full treatment cycle;
3. Patients with fungal, bacterial, viral or other uncontrollable infections or requiring four-level isolation treatment.
4. HIV, HBV and HCV positive;
5. Patients with diseases of the central nervous system or autoimmune central nervous system lesions, Including stroke, epilepsy, dementia;
6. Patients have myocardial infection, cardiac angiography or stents, active angina or other obvious clinical symptoms, or have cardiopathic asthma or cardiovascular lymphocytic infiltrates，within 12 months;
7. Patients are on anticoagulation or have severe coagulopathy (APTT>70);
8. Patients in any condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 2weeks prior to investigational drug administration;
9. Patients were infected with covid-19 within 2weeks prior to investigational drug administration;
10. Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator;
11. Subjects in other conditions that are considered unsuitable for this study by the investigator.-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Relief degree of tumors | through study completion, an average of 1 year
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST1.1）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 3 years, year 3
  The duration from the beginning of treatment to cancer recurrence or progression
Overall survival（OS） | 5 years, year 5
  The duration from the beginning of treatment to patient death

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China